CLINICAL TRIAL: NCT00434096
Title: A Randomized Double-blind, Placebo-controlled, Parallel-group, Fixed Single-dose Regimen (SR141716 20 mg), Multicenter Study to Assess the Efficacy and Safety of SR141716 in Obese Patients With Dyslipidemia.
Brief Title: Japanese Study of Rimonabant in Obese Patients With Dyslipidemia (VENUS)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision taken in light of demands by certain national health authorities
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC5749
Record Dates: First submitted 2007-02-09; First posted 2007-02-12 (Estimated); Last update posted 2009-07-20 (Estimated); Status verified 2009-07

CONDITIONS: Obesity
Keywords: Obesity disease; cannabinoid-1 receptor
MeSH Terms: conditions — Obesity | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: rimonabant (SR141716)
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: rimonabant (SR141716) — oral administration once daily
  Arms: 1
Drug: placebo — oral administration once daily
  Arms: 2

SUMMARY:
The primary objective of this study is to assess the efficacy of SR141716 compared to placebo on body weight and triglycerides changes over a period of 52 weeks.

Secondary objectives are:

* To evaluate the effect of SR141716 compared to placebo over a period of 52 weeks, on HDL-cholesterol and visceral fat area.
* To evaluate the safety of SR141716 compared to placebo over a period of 104 weeks.
* To evaluate the pharmacokinetics of SR141716.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) > 25 kg/m²
* Visceral Fat Area (VFA) > 100 cm²
* Triglycerides (TG) > 150 mg/dL and < 700 mg/dL, and/or HDL-cholesterol < 40 mg/dL(Dyslipidemia)
* At least 1 criteria of the following 2 comorbidities:

  * Impaired Glucose Tolerance or Type 2 diabetes
  * Hypertension

Exclusion Criteria:

* Patient with a secondary obesity.
* Patients who have received the diet therapy for less than 8 weeks before start of the observation period.
* Patients whose body weight changed by more than the variation of ± 2kg for screening period.
* Low compliance to drug intake (< 80%) and dietary instruction during the observation period.
* Patients with type 1 diabetes.
* Patients with a primary hyperlipidemia (i.e., familial hypercholesterolemia, familial combined hyperlipidemia and familial type III hyperlipidemia).
* Patients with a LDL-cholesterol > 190 mg/dL at any of Weeks -8 or -4.
* Patients with a secondary hypertension.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 915 (Actual)
Dates: Start 2007-02; Primary Completion 2008-11 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
body weight: relative change from baseline | Week 52
triglycerides: relative change from baseline | Week 52

SECONDARY OUTCOMES:
HDL-cholesterol ;visceral fat area | Week 52
Safety: Adverse events | study period

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Tokyo, Japan